CLINICAL TRIAL: NCT00435838
Title: A Retrospective, Multi-Centre Observational Study to Evaluate Disease Management and Adverse Events in Adult Subjects With HIV-1 Infection Who Were Withdrawn From CNA106030 Due to a Positive HLA-B*5701 Test Result
Brief Title: A Study of Patient Management in HIV-1 Infected Patients Found to Have the Genetic Marker HLA-B*5701
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Other Study IDs: CNA108223
Record Dates: First submitted 2007-02-15; First posted 2007-02-16 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: HIV Infection
Keywords: HLa-B*5701 Abacavir
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Retrospective

INTERVENTIONS:
Drug: No Intervention -- Observational study

SUMMARY:
This is a retrospective observational study which follows on from CNA106030 (a study evaluating whether prospective genetic screening for HLA-B*5701 can reduce the incidence of hypersensitivity reactions to abacavir). This study aims to collect data on approximately 35 subjects who withdrew from CNA106030 when found to be HLA-B*5701 positive. HIV disease management and adverse event data in these subjects, where the risk/benefit ratio of treatment with abacavir may alter subsequent prescribing, will be collected

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have received notification not to receive abacavir in the CNA106030 study because of a positive HLA-B*5701 screen result, and were subsequently withdrawn from protocol CNA106030.
* Subjects willing and able to understand and provide written informed consent prior to participation in this study.
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion criteria:

* Subjects who were not enrolled in the CNA106030 study
* Subjects who are not HLA-B*5701 positive
* Subjects who do not consent to being told their HLA-B*5701 status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 2007-03

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, PhD, Study Director — GlaxoSmithKline
Locations (23):
- Austria (4):
  - GSK Investigational Site, Graz
  - GSK Investigational Site, Innsbruck
  - GSK Investigational Site, Salzburg
  - GSK Investigational Site, Vienna
- GSK Investigational Site, Brussels, Belgium
- Italy (6):
  - GSK Investigational Site, Rimini, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Legnano (MI, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Bolzano, Trentino-Alto Adige
  - GSK Investigational Site, Padua, Veneto
- Russia (3):
  - GSK Investigational Site, Belgorod
  - GSK Investigational Site, Oryol
  - GSK Investigational Site, Volgograd
- GSK Investigational Site, Ljubljana, Slovenia
- Spain (7):
  - GSK Investigational Site, Alcalá de Henares
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Valencia
- GSK Investigational Site, La Chaux-de-Fonds, Switzerland